CLINICAL TRIAL: NCT01800214
Title: Prospective Neuroimaging, Cognition and Behavioural Study of Alzheimer's, Vascular, Parkinson's, Frontotemporal and Mixed Dementias
Brief Title: The Sunnybrook Dementia Study
Acronym: SDS
Status: Recruiting | Type: Observational
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: University of Toronto (Other); Sunnybrook Research Institute (Other); University of Waterloo (Other); Baycrest (Other)
Responsible Party: Principal Investigator, Dr. Sandra E Black, Brill Chair in Neurology, Sunnybrook Health Sciences Centre
Other Study IDs: CIHR MOP-13129; MOP-13129 (Other Grant/Funding Number: Canadian Institutes of Health Research)
Record Dates: First submitted 2013-02-25; First posted 2013-02-27 (Estimated); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Dementia
Keywords: neurodengeneration; neuroimaging
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood
  Retention: Samples with microbiome
  Description:
  Fecal Sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (8):
- Alzheimer's disease (AD)
- Vascular Cognitive Disorders (VCD)
- Lewy Body Disease (LBD)
- Frontotemporal Dementia (FTD): Behavioral-variant Frontotemporal Dementia (bvFTD) Language-variant Frontoemporal Dementia including Semantic dementia (SD) and Progressive non-fluent aphasia (PNFA) Corticobasal degeneration (CBD) Progressive supranuclear palsy (PSP)
- Mild Cognitive Impairment (MCI)
- Cognitively Normal (CN)
- Small Vessel Disease -Neurodegenerative (SVD)
- Subjective Cognitive Complaints (SCC)

SUMMARY:
The prospect of disease-modifying therapies in the pipeline for Alzheimer's Disease (AD) has intensified efforts to use brain imaging more effectively for diagnosis and monitoring of dementing illnesses. There is also emerging awareness of the destructive interplay between AD and Cerebrovascular Disease (CVD) in our aging population; both disorders share common vascular risk factors and may respond to similar prevention treatments. Brain mapping techniques capitalize on the fact that different neurodegenerative diseases target particular brain areas. Brain shrinkage and stroke disease can be quantified on Magnetic Resonance Imaging (MRI) using computerized analysis.

This ongoing study applies advanced MR imaging analysis, genetic testing and standardized cognitive and functional assessments done at yearly intervals to measure and monitor longitudinal change in patients with AD, vascular and other neurodegenerative diseases and potentially to measure modifying effects of emerging therapies. Over 1700 patients (Mild Cognitive Impairment or dementia from AD, Vascular, Frontotemporal or Lewy Body Disease) and 140 normal elderly have already been enrolled, with 180 autopsies.

This study utilizes specialized imaging analysis software packages to reliably quantify brain tissue volumes and small vessel disease, the most common type of CVD.

The SDS also investigates other potential biomarkers of dementia such as eye-tracking, optical coherence tomography, gait and balance, and the gut microbiome to explore their clinical utility.

Results from this study will help to improve diagnosis, to customize treatment, and to better monitor disease-modifying therapies currently under investigation should they become applicable to everyday practice.

ELIGIBILITY:
Patient Inclusion Criteria (General):

* Age between 40 and 90 (inclusive)
* Fluent in English
* Completed 8 years of education or higher
* Visual and auditory acuity adequate for neuropsychological testing
* Mini-Mental State Exam (MMSE) score ≥ 16

Patient Exclusion Criteria (General):

* Possible secondary causes of dementia, concomitant or history of neurological or psychiatric illness (other than stroke or Parkinsonism)
* History of alcohol or substance abuse or dependence within the past 2 years

Normal Control Inclusion Criteria:

* Age between 40-90
* Fluent in English
* Completed 8 years of education or higher
* No significant memory complaints

Normal Control Exclusion Criteria:

* Being treated or history of being treated for psychiatric or neurological illness
* History of alcohol or substance abuse or dependence within the past 2 years
* Current use of psychoactive medications (e.g. antidepressant, neuroleptics, chronic anxiolytics or sedative hypnotics, etc.)
* Medical contraindications to MRI

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population consisted of a sample of outpatients who attended a tertiary-care neurology clinic at the Sunnybrook Health Sciences Centre.
Sampling Method: Non-Probability Sample
Enrollment: 1800 (Estimated)
Dates: Start 1995-09; Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Volumetric change in brain structures and brain lesions on Magnetic Resonance Imaging (MRI) across the dementias covarying for age, sex, education and Apolipoprotein E (ApoE) status | 5 years
  Brain structures including whole brain, hippocampus, tissue volumes and cortical thickness in predefined regions of interest; brain lesions including lacunes, subcortical white matter hyperintensities, and stroke

SECONDARY OUTCOMES:
Rate of clinical decline as measured by detailed conventional neuropsychological testing, instrumental and standard activities of daily living assessments, caregiver forms, and behavioral psychiatric inventories | 5 years
Rate of change in perfusion patterns measured on Single Photon Emission Computerized Tomography (SPECT) at baseline and followup contrasts on a voxel-wise basis using Statistical Parametric Mapping (SPM), or in 79 predefined regions of interest | 5 years
Group differences for each cognitive, imaging and biomarker measurement | 5 years
Clinico-pathologic correlations between autopsy-confirmed histopathology and clinical features including clincial diagnosis, regaional atrophy, regional hypoperfusion, and white matter interintensities on MRI | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Sandra E Black, MD, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Callahan BL, Becker S, Ramirez J, Taylor R, Shammi P, Gao F, Black SE. Vascular Burden Moderates the Relationship Between ADHD and Cognition in Older Adults. Am J Geriatr Psychiatry. 2024 Apr;32(4):427-442. doi: 10.1016/j.jagp.2023.10.018. Epub 2023 Oct 30. PMID 37989710
- [Derived] Callahan BL, Ramakrishnan N, Shammi P, Bierstone D, Taylor R, Ozzoude M, Goubran M, Stuss DT, Black SE. Cognitive and Neuroimaging Profiles of Older Adults With Attention Deficit/Hyperactivity Disorder Presenting to a Memory Clinic. J Atten Disord. 2022 Jun;26(8):1118-1129. doi: 10.1177/10870547211060546. Epub 2021 Nov 16. PMID 34784815
- [Derived] Sapkota S, Ramirez J, Stuss DT, Masellis M, Black SE. Clinical dementia severity associated with ventricular size is differentially moderated by cognitive reserve in men and women. Alzheimers Res Ther. 2018 Sep 5;10(1):89. doi: 10.1186/s13195-018-0419-2. PMID 30185213
- [Derived] Saeed U, Mirza SS, MacIntosh BJ, Herrmann N, Keith J, Ramirez J, Nestor SM, Yu Q, Knight J, Swardfager W, Potkin SG, Rogaeva E, St George-Hyslop P, Black SE, Masellis M. APOE-epsilon4 associates with hippocampal volume, learning, and memory across the spectrum of Alzheimer's disease and dementia with Lewy bodies. Alzheimers Dement. 2018 Sep;14(9):1137-1147. doi: 10.1016/j.jalz.2018.04.005. Epub 2018 May 18. PMID 29782824
- [Derived] Swardfager W, Cogo-Moreira H, Masellis M, Ramirez J, Herrmann N, Edwards JD, Saleem M, Chan P, Yu D, Nestor SM, Scott CJM, Holmes MF, Sahlas DJ, Kiss A, Oh PI, Strother SC, Gao F, Stefanovic B, Keith J, Symons S, Swartz RH, Lanctot KL, Stuss DT, Black SE. The effect of white matter hyperintensities on verbal memory: Mediation by temporal lobe atrophy. Neurology. 2018 Feb 20;90(8):e673-e682. doi: 10.1212/WNL.0000000000004983. Epub 2018 Jan 26. PMID 29374101